CLINICAL TRIAL: NCT05302791
Title: Impact of Muscle Temperature on Muscle Growth and Breakdown: Cooling During Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0072-22-FB
Record Dates: First submitted 2022-03-07; First posted 2022-03-31 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Exercise Training
Keywords: Resistance Exercise; Muscle Cooling
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Each Subject acts as their own control in a de facto repeated measures design, where there is a Single bilateral exercise bout, with experimental and control assignment to individual limbs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Muscle Cooling (Experimental): The intervention will be applying a cooling wrap during the bilateral resistance exercise.
  Interventions: Device: Muscle Cooling; Other: Resistance Exercise
- Control (Placebo Comparator): There will be no temperature alteration for this leg during bilateral resistance exercise.
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Device: Muscle Cooling — Cooling wrap will be set to 10°C
  Arms: Muscle Cooling
Other: Resistance Exercise — Resistance Machines (Leg Press and Knee extension). 12 rep Max

SUMMARY:
The purpose of this study is to examine the effect of human skeletal muscle temperature during resistance exercise on myogenic and proteolytic signaling. Subjects will perform bilateral resistance exercise bouts at an intensity that should stimulate a muscle growth response in the Vastus Lateralis. During the resistance exercise, the subjects will receive a cold (10°C) intervention on the experimental limb, while receiving a neutral temperature intervention (22°C) on the control limb.

DETAILED DESCRIPTION:
A total of 2 visits to the laboratory will be required following the signing of informed consent. All visits will take place at the University of Nebraska Exercise Physiology Laboratory.

Initial Visit (~1.5-2 hours):

Height and weight will be measured using a medical scale. Body fat will be assessed with hydrostatic weighing using an electronic load cell based system (Exertech, Dresbach, MN) correcting for residual lung volume, or Bioelectrical Impedance Analysis body composition analyzer (InBodyUSA, Cerritos, CA) if needed.

Subjects will then perform a 12 Repetition (12RM) Max Test for bilateral seated leg press and seated leg extension using the following protocol on isotonic exercise machines at a weight designed to create failure between 8 and 12 repetitions. Following a short warm-up on a cycle ergometer, the subjects proceed with a bilateral leg press warm-up consisting of one set of ten repetitions at a self-determined light load, then one set of 5 repetition at a self-determined moderate load, and one set of 1 repetition at a predicted 12 rep maximum as predicted in relation to their Fat Free Mass. During the warm-up subjects will be coached on form, and observed for their ability to complete the repetition max test. Weight for the test will be altered to suit the subject's ability to complete approximately 12 repetitions. Once the desired weight is determined, subjects will be asked to complete as many repetitions as possible until the subject can no longer complete a repetition using a full range of motion. An identical testing protocol is then performed for the leg extension. This data will be used to estimate a 12RM workload, that would be appropriate for hypertrophic growth using the Watham equation .

Experimental Visit (~6.5-8 hours):

Participants will be instructed to arrive to the lab having fasted overnight, and they will be asked to avoid strenuous activity, alcohol consumption, tobacco use, and drug use for the 24 hour period leading up to experimental trial.

Subjects will complete the following experimental protocol briefly described: consume a small meal, a pre-exercise muscle biopsy, precool for 30 minutes, complete the exercise intervention, immediately post-exercise biopsy, 4 hour recovery with cooling, and post-recovery biopsy. At three time points (pre-exercise, immediately post-exercise, and post-4-hour recovery), skin temperature, muscle temperature, blood flow, and muscle tissue biopsies will be taken.

Details are as followed:

Meal When subjects arrive a consistent meal will be provided to standardize dietary intake. Food choices will be given to participants to create a meal between 700-800 calories, containing approximately 25-35 g of protein, 75-85 g of carbohydrates, and 35-45 g of fat. These foods will be made-up of commercially available pre-packaged foods. They will have approximately 30 minutes to consume their meal.

Cooling protocol Subjects will have Game Ready Med 4 elite thigh wraps around each thigh. This system circulates cooled liquid through a wrap specifically fitted for different body segments. One thigh will be cooled while the other thigh will be wrapped with the cuff, but not have any liquid circulating through it. These wraps do provide slight compression and thus it is important to apply the wraps to both legs. Each leg is assigned to either cold experimental group or control, will be randomized and counter-balanced between subjects. The liquid temperature circulating through the thermal wraps will be set to 10°C. The thermal wraps will be worn during a 30 minute cool down period prior to the exercise bout, during the exercise intervention, and during a 4 hour recovery period.

Exercise Intervention The subjects will complete an intervention designed to stimulate the muscle growth signaling pathway (hypertrophy) in the Vastus Lateralis (outer thigh), via bilateral seated leg press and bilateral seated leg extension on isotonic exercise machines. Subjects will perform four sets of bilateral leg press exercises at the weight determined to be their 12 RM from the repetition max test. This should allow completion to failure of 8-12 repetitions. So, if more than 12 reps are able to be completed, weight will be added to the resistance for the subsequent sets. Conversely, if less than 8 reps lead to failure, the weight should be reduced for the subsequent sets. Constant dialogue with subjects will give investigators the ability to monitor set weights to maximize a hypertrophic response. Subjects will be allowed 2 minute of rest between each set. Upon completion of 4 sets, the subjects will be given 5 minutes of rest prior to repeating this protocol for bilateral leg extensions.

Biopsies A total of 6 muscle biopsies (1 per leg) will be obtained from the vastus lateralis (outer thigh) muscle. One from each leg for each of the 3 collection time-points, pre-exercise, immediately post-exercise, and post-4-hour recovery. Briefly, the area above the vastus lateralis muscle belly will be shaved and cleaned with alcohol. 1% xylocaine is then injected under the skin with a 25 ga hypodermic needle. The area is then further disinfected with betadine, and a sterile fenestrated drape is placed over the biopsy site. Using sterile techniques, a small incision is made through the skin (~5mm) and the Bergstrom biopsy needle is inserted through the incision into the belly of the muscle. The Bergstrom needle then takes a small clip of muscle (~50mg) and is removed from the muscle and stored in a chemical stabilizer. Slight pressure is held over the incision for approximately 2 minutes and is then closed using steri-strips and a band-aid with antibiotic ointment.

Intramuscular Temperature Using the incision from the muscle biopsy, a hypodermic (~26ga) thermocouple (Physitemp Instruments LLC, Clifton, NJ) that is smaller than the needle used to inject the xylocaine will be inserted into the belly of the muscle to measure intramuscular temperature. The thermocouple readings stabilize in approximately 3 seconds and the thermocouple is then removed. Recordings for intramuscular temperature will be collected during the biopsy process following the intervention.

Skin Temperature Skin Temperature will be measured on the surface of each thigh using a skin thermistor (Physitemp Instruments LLC, Clifton, NJ), infrared digital thermometer, and/or using an infrared thermal camera. Measurements will be taken at the same time as the intramuscular. The thermistor is simply placed on the skin for approximately 3 seconds and is then recorded. The infrared thermal camera can measure and record surface temperatures for a field of multiple surfaces.

ELIGIBILITY:
Inclusion Criteria:

* Any male or female who is 19-45 of age and is considered
* low risk for physical activity based on the American College of Sports Medicine (ACSM) guidelines
* recreationally active during the 6 weeks prior to participation by meeting the ACSM minimum activity guidelines

Exclusion Criteria:

* Any person outside of the age range of 19-45
* not considered 'low risk' on the ACSM Risk Stratification Form
* not meeting the exercise requirements for the preceding 6 weeks will be excluded.
* self-report of a history of joint or muscular injury that would prevent them from safely completing the required activities
* self-report of taking prescription drugs or supplements that may interfere with this research
* self-report allergy to Xylocaine
* pregnant
* breast feeding
* self-report sensitivity to heat or cold

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin R Slivka, PHD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: experimental (cooling) or control
Groups:
- All Participants: all participants have one leg serving as the experimental (10 degrees C cooling wrap) and the other as the control (no cooling) before, during, and after resistance exercise.
Period: Overall Study
Arm/Group | All Participants
Started | 12; 24 experimental (cooling) or control
Experimental (Cooling) | 12; 12 experimental (cooling) or control
Control (no Cooling) | 12; 12 experimental (cooling) or control
Completed | 12; 24 experimental (cooling) or control
Not Completed | 0; 0 experimental (cooling) or control

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12
height [Mean (Standard Deviation); unit: meters] | 1.71 (.08)
weight [Mean (Standard Deviation); unit: kg] | 77.3 (15.9)
body composition [Mean (Standard Deviation); unit: % fat] | 20.8 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: RT-qPCR for Forkhead Box O3 (FOXO3a)
Description: RT-qPCR for Forkhead Box O3 (FOXO3a) [mRNA response FOXO3a]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 1.24 (.69) | 1.30 (.98)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .609, ANOVA; time x condition ANOVA

2. Primary Outcome: RT-qPCR for Tripartite Motif Containing 63 (TRIM63)
Description: RT-qPCR for Tripartite Motif Containing 63 (TRIM63) [mRNA response of TRIM63]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 3.59 (3.4) | 3.50 (4.43)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .858, ANOVA; time x condition anova

3. Primary Outcome: RT-qPCR for Growth/Differentiation Factor 8 (MSTN)
Description: RT-qPCR for Growth/Differentiation Factor 8 (MSTN) [mRNA response of MSTN]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | .44 (.3) | .44 (.29)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .633, ANOVA

4. Primary Outcome: RT-qPCR for Myogenic Factor 5 (MYF5)
Description: RT-qPCR for Myogenic Factor 5 (MYF5) [mRNA response of MYF5]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | .51 (.21) | .83 (.55)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .076, ANOVA

5. Primary Outcome: RT-qPCR for Myogenic Factor 6 (MYF6)
Description: RT-qPCR for Myogenic Factor 6 (MYF6) [mRNA response of MYF6]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 2.2 (1.7) | 1.32 (.47)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .151, ANOVA

6. Primary Outcome: RT-qPCR for Myocyte Enhancer Factor 2A (MEF2a)
Description: RT-qPCR for Myocyte Enhancer Factor 2A (MEF2a) [mRNA response of MEF2a]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 1.44 (1.28) | 1.91 (2.12)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .385, ANOVA

7. Primary Outcome: RT-qPCR for Myogenic Differentiation 1 (MYOD1)
Description: RT-qPCR for Myogenic Differentiation 1 (MYOD1) [mRNA response of MYOD1]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 2.08 (1.73) | 1.92 (1.6)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .665, ANOVA

8. Primary Outcome: RT-qPCR for Myogenin (MYOG)
Description: RT-qPCR for Myogenin (MYOG) [mRNA response of MYOG]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 1.88 (1.75) | 2.62 (1.33)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .078, ANOVA

9. Primary Outcome: RT-qPCR for Ribosomal Protein S3 (RPS3)
Description: RT-qPCR for Ribosomal Protein S3 (RPS3) [mRNA response of RPS3]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 1.46 (1.55) | 1.29 (.69)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .773, ANOVA

10. Primary Outcome: RT-qPCR for Ribosomal Protein L3 Like (RPL3L)
Description: RT-qPCR for Ribosomal Protein L3 Like (RPL3L) [mRNA response of RPL3L]
  Fold change calculated using the delta, delta CT method relative to stable reference genes and pre-exercise measures.
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: fold change
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
fold change | 1.55 (1.57) | .78 (.34)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p = .118, ANOVA

11. Secondary Outcome: Muscle Temperature
Description: Intramuscular Temperature
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: degrees C
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
degrees C | 26.09 (3) | 35.07 (1.04)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p < 0.001, ANOVA; Time x condition ANOVA

12. Secondary Outcome: Skin Temperature
Description: Surface Temperature of the skin
Time Frame: 4-hours post Exercise
Measure: Mean (Standard Deviation); unit: degrees C
Units Other Than Participants: legs
Arm/Group | Muscle Cooling | Control
Number analyzed (Participants) | 12 | 12
Number analyzed (legs) | 12 | 12
degrees C | 20.4 (2.01) | 31.65 (2.04)
Statistical Analysis 1: Comparison: Muscle Cooling vs Control; Test type: Superiority; p < 0.001, ANOVA; time x condition anova

ADVERSE EVENTS:
Time Frame: adverse event data was collected from initial visit to the completion of the study for each participant, approximately 2 months.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT05302791/Prot_SAP_000.pdf